CLINICAL TRIAL: NCT05818657
Title: Prevalence of of Apical Periodontal in Patients Chronic Kidney Disease & Its Association With Markers of Kidney Disease.
Brief Title: Association of Apical Periodontitis With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Dr. Jyoti Lamba
Record Dates: First submitted 2021-12-11; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Diseases; Periapical Lesions
Keywords: Apical Periodontitis; Root Canal Treatment
MeSH Terms: conditions — Renal Insufficiency, Chronic; Periapical Periodontitis | interventions — Health Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood analysis for CRP, Serum ferritin, Albumin, Creatinine & Urea
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-A CKD patients: Prevalence of apical periodontitis will be checked and non-surgical root canal treatment will be given to the patients with apical periodontitis and change in PAI score, eGFR & Systemic markers will be checked
  Interventions: Biological: levels of CKD markers, Oral health status, apical periodontitis
- Group-B Healthy individuals: Prevalence of apical periodontitis will be checked and non-surgical root canal treatment will be given to the patients with apical periodontitis and change in PAI score, eGFR & Systemic markers will be checked
  Interventions: Biological: systemic inflammatory marker, Oral health status, apical periodontitis

INTERVENTIONS:
Biological: levels of CKD markers, Oral health status, apical periodontitis — To observe levels of CKD markers :Levels of serum keratinise ,urea, eGFR, and assessment of Oral health status, apical periodontitis
  Groups: Group-A CKD patients
Biological: systemic inflammatory marker, Oral health status, apical periodontitis — estimation of hs-CRP levels, and assessment of Oral health status, apical periodontitis
  Groups: Group-B Healthy individuals

SUMMARY:
This investigation is aimed to assess the prevalence and severity of apical periodontitis (AP) in different stages of CKD patients and its impact on the systemic (nutritional and inflammatory) markers was compared to healthy individuals.

DETAILED DESCRIPTION:
105 CKD patients (35 early (EG), 35pre-dialysis (PDG) and 35 hemodialysis (HDG)groups and 105 age and gender matched healthy controls were assessed for prevalence and severity of apical periodontitis and oral disease burden . Inflammatory (hsCRP and ferritin) and nutritional (urea and creatinine) markers were estimated and eGFR was calculated for the study population. Logistic regression was used to determine the possible association between CKD and AP in study population and Linear regression was performed to evaluate the possible association between systemic markers and endodontic burden (EB) in experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Known patient of CKD Stages 1,2,3,4 & 5 with estimated glomerular filtration rate [eGFR; MDRD] with mature permanent teeth.
* > 18 years
* > 8 natural teeth.
* Complete medical & dental history including panoramic radiographs of maxilla & mandible

Exclusion Criteria:

* Patients having systemic disorders other than CKD (eg HIV, Diabetes mellitus, Coronary heart disease, history of secondary hyperparathyroidism).
* Pregnancy, lactation & contraceptives.
* Systemic conditions that contra indicates dental treatment.
* Use of antibiotics & anti-inflammatory in last 3 months
* Need for antibiotic prophylaxis.
* Hepatitis C and B virus.
* Patients on steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD patients of different levels (Stage 1 to Stage 5) with age and gender matched controls will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Periapical Index(PAI) | 1 year
  Periodical status will be assessed in periodical radiograph and scoring of periapical index will be done according to size and periphery of peri-apical radiolucency with coding 1 to 5
eGFR | 1 year
  BY BLOOD SAMPLE measured in mL/min/1.73m2
serum creatinine | 1 year
  BY BLOOD SAMPLE measured in mg/dL
hs-CRP | 1 year
  HIGH SENSITIVE C-reactive protein measured by ELISA kit in mg/L
Blood urea | 1 year
  measured by collecting blood sample in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shweta Mittal, MDS, Study Director — Post Graduate Institute Of Dental Sciences, Rohtak.
Locations (1):
- PGIDS, Rohtak, Haryana, India